CLINICAL TRIAL: NCT02067728
Title: Family Nutrition, Physical Activity (FNPA) Tool: a Motivational Interviewing-based Practice Intervention to Address Pediatric Health Behaviors
Brief Title: Family Nutrition Physical Activity Tool Use During Well Child Visits
Acronym: FNPA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: American Cancer Society, Inc. (Other); Northwestern University Feinberg School of Medicine (Other); New York University (Other)
Responsible Party: Principal Investigator, Amy Christison, M.D., Clinical Assistant Professor, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 297832
Record Dates: First submitted 2014-02-16; First posted 2014-02-20 (Estimated); Results first posted 2016-03-23 (Estimated); Last update posted 2016-03-23 (Estimated); Status verified 2016-02

CONDITIONS: Obesity
Keywords: obesity prevention
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Usual Care (Active Comparator): Usual care is provided to patients in practice groups not undergoing intervention of FNPA tool
  Interventions: Behavioral: Usual Care
- FNPA tool intervention (Experimental): FNPA tool practice intervention comprising of two components: 1) FNPA assessment which screens for obesigenic behaviors; 2) Brief Action Planning conversation designed to assist the family develop a health behavior change goal based on obesigenic risks on the assessment tool.
  Interventions: Behavioral: FNPA tool

INTERVENTIONS:
Behavioral: FNPA tool — Intervention practice will train to use FNPA screening paired with Brief Action Planning. They will implement this approach during well child visits.
  Arms: FNPA tool intervention
Behavioral: Usual Care — Practices not undergoing intervention with FNPA tool will provide usual care to patients during well-child visits.
  Arms: Usual Care

SUMMARY:
The main aim of the study would be to examine the effect of using a health behavior screening tool and a brief patient centered conversation on health behavior goal setting during well-child visits.

DETAILED DESCRIPTION:
Rationale and Significance: Although much research aimed at preventing childhood obesity focuses on community, environment, and school-based initiatives, there is significant potential for healthcare systems and primary care providers to aid in preventing obesity. All children, one-third of whom are overweight, have multiple well-child and acute encounters with their providers. Provider counseling regarding Body Mass Index (BMI) is strongly correlated with a parent's perception of his or her child's weight, and parents who perceive BMI as a health problem are 10 times more likely to make healthy lifestyle changes.As a result, a practice intervention aimed at improving behavior change goals employed during well-child encounters provide an optimal opportunity for physicians to impact family lifestyle behaviors and hopefully reduce the trajectory of obesity rates in their patient population.

To our knowledge, there is little published evidence regarding the use of validated, brief, screening and coaching tools paired with MI-enhanced conversations related to obesigenic behaviors during health supervision visits. The proposed project, a practice-based intervention that pairs Brief Action Planning (BAP)focused on targeted obesigenic behaviors identified by the Family Nutrition Physical Activity (FNPA ) tool, addresses many of the barriers of existing current practice approaches and will enable providers to implement a focused conversation to establish realistic behavior change goals. The study brings primary care providers to the forefront of obesity prevention while allowing the patient to direct the path to behavior change. The intervention includes a patient-centered approach and has been proven to be feasible and acceptable among providers and patients. The potential impact of this project is to increase provider and patient collaboration for goal-setting, which will then result in a reduction of obesigenic behaviors. Evidence from this investigation will give providers specific and feasible methods for counseling on behaviors associated with obesity.

Procedures:

Practice Recruitment: For 3 months, practice recruitment meetings will be held with offices from three healthcare networks during which the research protocol will be explained, roles and responsibilities of research staff and practices will be outlined, and written agreements signed. At baseline, all practices will complete a practice and provider demographic questionnaire to characterize any baseline procedures and documentation practices related to obesity prevention as well as previous provider training in obesity prevention and MI (questionnaire is available on request). Practices will then be matched and randomly assigned.

Practice training: Practitioners will have a four-month period to undergo three 1.5-hour training sessions to learn the principles of MI and BAP and get familiar with using the FNPA tool. Research staff and trainers who are licensed clinical professional counselors (LCPC) certified in BAP will lead trainings. A PhD psychologist researcher will develop the curriculum and oversee trainers. Competency will be measured by successful certification of a BAP encounter and correctly interpreting three FNPA tools. Trained research staff will teach office staff correct techniques in anthropometrics and FNPA scoring. Competency will be measured by three accurate measurements and correct scoring of three FNPA tools. Scales and stadiometers at each enrolled practice will be calibrated for consistency in measurement across sites.

Subject Recruitment: Subject recruitment will occur one month before implementation. Eligible subjects with scheduled well-child visits will receive a letter signed by their provider and the PI (Amy Christison, MD). The letter will briefly describe the study and offer the opportunity to enroll. They will be given an opt-out phone number to call within one week of mailing this letter if they do not want to participate. If the research coordinator does not receive a call, he/she will contact the family by phone to answer questions and send a consent form to the family. The subject will be considered enrolled after obtaining a signed written consent from the family.

Implementation Period: The FNPA tool will be routinely used during all health supervision visits in the implementation practices during 6 months, regardless of patient is enrolled or not. During scheduled well child visits, treatment group practices will implement the FNPA tool using BAP. Parents/guardians of all patients, ages 4 to 11, will be asked to answer the FNPA child questionnaire, and patients, ages 12 to 17, with their parents will answer the FNPA adolescent questionnaire. The practice staff will score it, and providers will 1) engage the family in a patient-centered discussion about the patient's body mass index (BMI) percentage ,2) discuss healthy and obesigenic behaviors identified on the tool, 3) mutually decide on any goals for change, 4) determine the patient's confidence for change, and 5) offer follow-up by phone or appointment regarding stated goals, and 6) offer follow-up appointments for focused counseling of patients identified as overweight or obese as per American Academy of Pediatrics (AAP) recommendations. Goals and follow-up plans will be documented on the FNPA tool, and copies will be given to the family and retained in the chart. For healthy weight children, if follow-up by phone call is chosen, it will be implemented at the time selected by the patient and by the clinical research staff trained in BAP so that lack of support staff in a particular site for such calls is not a confounding variable.

Control group practices will provide usual well-child care per AAP recommendations.Their patients will complete an FNPA assessment questionnaire directly after their appointment for the purposes of comparing baseline and end point measures. Importantly, this approach prevents the possibility of providers commenting on the results.

Both treatment and control group parents/guardians of patients attending appointments will provide demographic data including parent-reported parent weight and height, and income range. Age, sex, and patient calculated BMI and z-score will be abstracted from the medical record.

Outcomes Measurement Procedures:

1. Treatment group patients will rate their impressions of the FNPA tool at the end of the appointment. If patients are adolescents (12 years or older), both the patient and the attending parent will complete the survey. Parents of younger children will complete surveys for those patients.
2. A research assistant blinded to treatment group will perform all phone surveys. At 1 month, patients from both groups will be will be asked to rate how patient centered their encounter was. Behavior change surveys will be performed at 1 month and 6 months following the encounter.
3. All subjects will be asked to return to their practices for weight and height measurements 6 months after their initial encounter and to fill out a second FNPA tool. This will be performed by un-blinded research staff as using blinding in this setting would not be feasible.
4. Audit of charting regarding goal setting documentation, successful identification of overweight and obese patients, and compliance with recommended follow-up appointments will be performed of both groups.
5. Treatment group providers will have a baseline and two random encounters audio recorded midway and at the end of the intervention period. They will be scored for fidelity to the BAP-approach by a trained and blinded coder. This is done to understand the effectiveness of the BAP training for the provider. They will also receive feedback from the coding results and given a refresher if needed. Control group providers will have one baseline encounter recorded and scored for fidelity and comparison to treatment group providers.
6. Providers will be surveyed regarding their satisfaction with the FNPA intervention at the end of the 6-month intervention time.

Analysis: Analysis will be done with Statistical Analysis System (SAS) 9.3 or the latest version. A significance level of p<=0.05 is accepted as significant. Descriptive statistics (mean, median, mode, range) will be examined and the data set cleaned. To compare the two study groups for univariate analysis, t-tests will be computed for interval variables, Mann-Whitney U for ordinal variables, and Chi-square for nominal variables. Generalized Linear Mixed Models will be employed for multivariate analysis with repeated measures and multi-level effects. Subjects who drop out or are lost to follow-up will be compared to completed subjects in differences related to demographics, socioeconomic status, and BMI.

ELIGIBILITY:
Inclusion Criteria:

- All children ages 4-17 years scheduled for well child visits

Exclusion Criteria:

-Patients with chronic medical conditions or developmental delays that preclude age appropriate nutrition and physical activity habits will be excluded. -

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 430 (Actual)
Dates: Start 2014-02; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amy Christison, MD, Principal Investigator — University of Illinois College of Medicine at Peoria
Locations (1):
- UnityPointHealth Methodist in Peoria, Peoria, Illinois, United States

REFERENCES:
- [Background] Campbell K, Waters E, O'Meara S, Summerbell C. Interventions for preventing obesity in children. Cochrane Database Syst Rev. 2001;(3):CD001871. doi: 10.1002/14651858.CD001871. PMID 11686999
- [Background] Gutnick D. Brief Action Planning to Facilitate Behavior Change and Support Patient Self-Management.Journal of Clinical Outcomes Management 21(1):17-29, 2014
- [Background] Taveras EM, Gortmaker SL, Hohman KH, Horan CM, Kleinman KP, Mitchell K, Price S, Prosser LA, Rifas-Shiman SL, Gillman MW. Randomized controlled trial to improve primary care to prevent and manage childhood obesity: the High Five for Kids study. Arch Pediatr Adolesc Med. 2011 Aug;165(8):714-22. doi: 10.1001/archpediatrics.2011.44. Epub 2011 Apr 4. PMID 21464376
- [Background] Barlow SE; Expert Committee. Expert committee recommendations regarding the prevention, assessment, and treatment of child and adolescent overweight and obesity: summary report. Pediatrics. 2007 Dec;120 Suppl 4:S164-92. doi: 10.1542/peds.2007-2329C. PMID 18055651
- [Background] Huang JS, Donohue M, Golnari G, Fernandez S, Walker-Gallego E, Galvan K, Briones C, Tamai J, Becerra K. Pediatricians' weight assessment and obesity management practices. BMC Pediatr. 2009 Mar 5;9:19. doi: 10.1186/1471-2431-9-19. PMID 19265553
- [Background] Perrin EM, Flower KB, Garrett J, Ammerman AS. Preventing and treating obesity: pediatricians' self-efficacy, barriers, resources, and advocacy. Ambul Pediatr. 2005 May-Jun;5(3):150-6. doi: 10.1367/A04-104R.1. PMID 15913408
- [Background] Story MT, Neumark-Stzainer DR, Sherwood NE, Holt K, Sofka D, Trowbridge FL, Barlow SE. Management of child and adolescent obesity: attitudes, barriers, skills, and training needs among health care professionals. Pediatrics. 2002 Jul;110(1 Pt 2):210-4. PMID 12093997
- [Background] Berg-Smith SM, Stevens VJ, Brown KM, Van Horn L, Gernhofer N, Peters E, Greenberg R, Snetselaar L, Ahrens L, Smith K. A brief motivational intervention to improve dietary adherence in adolescents. The Dietary Intervention Study in Children (DISC) Research Group. Health Educ Res. 1999 Jun;14(3):399-410. doi: 10.1093/her/14.3.399. PMID 10539230
- [Background] Erickson SJ, Gerstle M, Feldstein SW. Brief interventions and motivational interviewing with children, adolescents, and their parents in pediatric health care settings: a review. Arch Pediatr Adolesc Med. 2005 Dec;159(12):1173-80. doi: 10.1001/archpedi.159.12.1173. No abstract available. PMID 16330743
- [Background] Taveras EM, Mitchell K, Gortmaker SL. Parental confidence in making overweight-related behavior changes. Pediatrics. 2009 Jul;124(1):151-8. doi: 10.1542/peds.2008-2892. PMID 19564295
- [Background] Schwartz RP, Hamre R, Dietz WH, Wasserman RC, Slora EJ, Myers EF, Sullivan S, Rockett H, Thoma KA, Dumitru G, Resnicow KA. Office-based motivational interviewing to prevent childhood obesity: a feasibility study. Arch Pediatr Adolesc Med. 2007 May;161(5):495-501. doi: 10.1001/archpedi.161.5.495. PMID 17485627
- [Background] Bodenheimer T, Handley MA. Goal-setting for behavior change in primary care: an exploration and status report. Patient Educ Couns. 2009 Aug;76(2):174-80. doi: 10.1016/j.pec.2009.06.001. Epub 2009 Jun 27. PMID 19560895
- [Background] Shilts MK, Horowitz M, Townsend MS. Goal setting as a strategy for dietary and physical activity behavior change: a review of the literature. Am J Health Promot. 2004 Nov-Dec;19(2):81-93. doi: 10.4278/0890-1171-19.2.81. PMID 15559708
- [Background] Gans KM, Ross E, Barner CW, Wylie-Rosett J, McMurray J, Eaton C. REAP and WAVE: new tools to rapidly assess/discuss nutrition with patients. J Nutr. 2003 Feb;133(2):556S-62S. doi: 10.1093/jn/133.2.556S. PMID 12566502
- [Background] Patrick K, Sallis JF, Prochaska JJ, Lydston DD, Calfas KJ, Zabinski MF, Wilfley DE, Saelens BE, Brown DR. A multicomponent program for nutrition and physical activity change in primary care: PACE+ for adolescents. Arch Pediatr Adolesc Med. 2001 Aug;155(8):940-6. doi: 10.1001/archpedi.155.8.940. PMID 11483123
- [Background] Ihmels MA, Welk GJ, Eisenmann JC, Nusser SM. Development and preliminary validation of a Family Nutrition and Physical Activity (FNPA) screening tool. Int J Behav Nutr Phys Act. 2009 Mar 12;6:14. doi: 10.1186/1479-5868-6-14. PMID 19284631
- [Background] Ihmels MA, Welk GJ, Eisenmann JC, Nusser SM, Myers EF. Prediction of BMI change in young children with the family nutrition and physical activity (FNPA) screening tool. Ann Behav Med. 2009 Aug;38(1):60-8. doi: 10.1007/s12160-009-9126-3. Epub 2009 Oct 6. PMID 19806417

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a randomized controlled trial comprised of 12 primary care clinics within the Peoria, Illinois region, providing well-child care to children ages 4-17 years. Clinics were a combination of pediatric, medicine/pediatric, and family medicine clinics. Study group assignments were determined by size, specialty, and socioeconomic demographics.
Pre-assignment Details: Practices were paired and then randomized to assure similarity across intervention and usual care groups. A total of 35 Providers participated and 430 children/family were enrolled into the project.
Period: Baseline - 1 Month Follow up Survey
Arm/Group | Usual Care | FNPA Tool Intervention
Started | 220 | 210
Completed | 213 (213 parents/guardians completed the surveys, along with 82 teens.) | 182 (182 parent/guardians completed the surveys, along with 75 teens.)
Not Completed | 7 | 28
Not completed — Lost to Follow-up | 7 | 28
Period: 6 Month Follow up Survey
Arm/Group | Usual Care | FNPA Tool Intervention
Started | 220 (Participants completed the 6 month follow up even if 1 month data wasn't able to be collected.) | 210 (Participants completed the 6 month follow up even if 1 month data wasn't able to be collected.)
Completed | 172 (172 parent/guardians completed surveys at this time point, along with 71 teens.) | 150 (150 parent/guardians completed surveys at this time point, along with 69 teens.)
Not Completed | 48 | 60
Not completed — Lost to Follow-up | 48 | 60
Period: 6 Month Measurements
Arm/Group | Usual Care | FNPA Tool Intervention
Started | 220 | 210
Completed | 106 (Number includes 6 month measurements & chart review for visits at 6 months +/- 2 months from initial) | 113 (Number includes 6 month measurements & chart review for visits at 6 months +/- 2 months from initial)
Not Completed | 114 | 97
Not completed — Unable to attend | 114 | 97

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | FNPA Tool Intervention | Total
Number analyzed (Participants) | 220 | 210 | 430
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 220 | 210 | 430
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.4 (4.1) | 10.7 (4.1) | 10.6 (4.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 113 | 117 | 230
  Male | 107 | 93 | 200
Region of Enrollment [Number; unit: participants]
  United States | 220 | 210 | 430
Body Mass Index [Mean (Standard Deviation); unit: kg/m²] | 19.8 (5.1) | 20.0 (5.0) | 19.9 (5.1)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With Documented Goal Setting
Description: Health behavior change goal documented in charting of well-child visits.
Time Frame: 2 weeks from encounter
Population: Manual chart review of the electronic medical record (EMR) was completed by the Research Team for all enrolled subjects in both study groups. Goal documentation was defined as any type of goal consisting of an active verb written either on the FNPA Tool which was completed during the well child visit or in Physician notes in the EMR for the visit.
Measure: Number; unit: percentage of participant charts
Arm/Group | Usual Care | FNPA Tool Intervention
Number analyzed (Participants) | 220 | 210
percentage of participant charts | 4.09 | 71.90

2. Secondary Outcome: Obesiogenic Goal Setting Success
Description: Degree to which an obesiogenic goal was set and carried out at 1 month after the encounter. Success defined as response of 2-4 on health behaviors survey, with 2=success some of the time, 3=success most of the time, and 4=success almost always.
Time Frame: 1 month after the encounter
Population: This analysis population only includes the participants who set an obesiogenic goal at the initial appointment and completed the 1 month post survey to rate their success level in achieving that goal.
Measure: Number; unit: percentage of participants
Arm/Group | Usual Care | FNPA Tool Intervention
Number analyzed (Participants) | 55 | 138
percentage of participants | 87.27 | 98.55
Statistical Analysis 1: Comparison: Usual Care vs FNPA Tool Intervention; Test type: Superiority or Other; p = 0.0029, Chi-squared

3. Other Pre Specified Outcome: BMI Z-score Change for All
Description: Anthropometric measures of weight and height and calculated BMI z score change at 6 months post encounter.
Time Frame: Baseline and 6 months after the encounter
Population: The number of participants analyzed is low because returning for measurement checks was optional at 6 months & only 28% usual care and 27% intervention group attended. We also included chart abstraction measurements for those who had a return clinic visit with measurements within 6 months +/- 2 months from initial encounter.
Measure: Mean (Standard Deviation); unit: BMI z-score
Arm/Group | Usual Care | FNPA Tool Intervention
Number analyzed (Participants) | 106 | 113
BMI z-score | 0.14 (0.51) | 0.08 (0.42)
Statistical Analysis 1: Comparison: Usual Care vs FNPA Tool Intervention; Test type: Superiority or Other; p = 0.3875, t-test, 2 sided

4. Other Pre Specified Outcome: Perception of Patient Centeredness of Encounter
Description: Patient centeredness survey which measures the parent's and patient's (if 12 years and older) perception of how patient centered the communication was with the provider. Survey Coding for Patient Centeredness: 1=Not at all; 2=A little; 2.5=Can't say; 3=Somewhat; 4=A lot
Time Frame: 1 month after the encounter
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Care | FNPA Tool Intervention
Number analyzed (Participants) | 193 | 179
units on a scale | 3.42 (0.45) | 3.67 (0.39)
Statistical Analysis 1: Comparison: Usual Care vs FNPA Tool Intervention; Test type: Superiority or Other; p < 0.05, t-test, 2 sided; Mean Difference (Net) = -0.26, Standard Deviation 0.42

5. Other Pre Specified Outcome: Obesity Follow-up Adherence
Description: Subjects identified as obese with recommended follow-up appointment who are adherent to recommendation within 6 months of encounter
Time Frame: 6 months after the encounter
Population: This analysis population only includes the subjects who were identified as obese at their initial appointment and had a 6 month follow up appointment scheduled at that time.
Measure: Number; unit: percentage of participants
Arm/Group | Usual Care | FNPA Tool Intervention
Number analyzed (Participants) | 4 | 2
percentage of participants | 50 | 50
Statistical Analysis 1: Comparison: Usual Care vs FNPA Tool Intervention; Test type: Superiority or Other; p > 0.05, Chi-squared

6. Secondary Outcome: Obesiogenic Goal Setting Success
Description: Degree to which an obesiogenic goal was set and carried out at 6 months after the encounter. Success defined as response of 2-4 on survey, with 2=success some of the time, 3=success most of the time, and 4=success almost always.
Time Frame: 6 months after encounter
Population: This analysis population only includes the subjects who had initially set an obesiogenic goal at the well child appointment and responded to the survey at 6 months after the medical encounter when goal was set.
Measure: Number; unit: percentage of participants
Arm/Group | Usual Care | FNPA Tool Intervention
Number analyzed (Participants) | 50 | 121
percentage of participants | 100 | 99.17
Statistical Analysis 1: Comparison: Usual Care vs FNPA Tool Intervention; Test type: Superiority or Other; p = 1.000, Chi-squared

7. Secondary Outcome: Success of Obesiogenic Goals
Description: Degree to which an obesiogenic goal was set and successfully carried out at 1 month post encounter. Success is defined as rating of 3 or 4 on the 1 month health behavior survey, with 3=goal met most of the time and 4= goal met almost always.
Time Frame: 1 month post encounter
Population: This analysis population only includes the subjects who had initially set an obesiogenic goal at the well child appointment and responded to the survey at 1 month after the medical encounter to rate their level of success in achieving that goal.
Measure: Number; unit: percentage of participants
Arm/Group | Usual Care | FNPA Tool Intervention
Number analyzed (Participants) | 210 | 178
percentage of participants | 17.14 | 56.18
Statistical Analysis 1: Comparison: Usual Care vs FNPA Tool Intervention; Test type: Superiority or Other; p < 0.0001, Chi-squared; Risk Ratio (RR) = 3.3, 95% CI 2-sided [2.2 to 4.9]

8. Secondary Outcome: Success of Obesiogenic Goals
Description: Degree to which an obesiogenic goal was set and successfully carried out at 6 months post encounter. Success is defined as rating of 3 or 4 on the 1 month health behavior survey, with 3=goal met most of the time and 4= goal met almost always.
Time Frame: 6 months post encounter
Population: This analysis population only includes those participants who initially set an obesiogenic focused goal at their well child check and then responded to the survey 6 months after to rate their success level in achieving that goal.
Measure: Number; unit: percentage of participants
Arm/Group | Usual Care | FNPA Tool Intervention
Number analyzed (Participants) | 170 | 150
percentage of participants | 20.59 | 60.67
Statistical Analysis 1: Comparison: Usual Care vs FNPA Tool Intervention; Test type: Superiority or Other; p < 0.0001, Chi-squared; Risk Ratio (RR) = 2.9, 95% CI 2-sided [2.0 to 4.5]

9. Secondary Outcome: Success of Other Health Goals
Description: Degree to which other health behavior goals (non-obesiogenic) were set and carried out at 1 month post encounter. Success defined as response of 2-4 on health behaviors survey, with 2=success some of the time, 3=success most of the time, and 4=success almost always.
Time Frame: 1 month post encounter
Population: This analysis population only includes subjects who set a health goal, which was not obesiogenic focused, during the initial visit and responded to the survey regarding success of achieving the goal 1 month post encounter.
Measure: Number; unit: percentage of participants
Arm/Group | Usual Care | FNPA Tool Intervention
Number analyzed (Participants) | 26 | 33
percentage of participants | 88.46 | 90.91

10. Secondary Outcome: Success of Other Health Goals
Description: Degree to which other health behavior goals (non-obesiogenic) were set and carried out at 6 months post encounter. Success defined as response of 2-4 on health behaviors survey, with 2=success some of the time, 3=success most of the time, and 4=success almost always.
Time Frame: 6 months post encounter
Population: This analysis population only includes subjects who set a health goal, which was not obesiogenic focused, during the initial visit and responded to the survey regarding success of achieving the goal 6 months post encounter.
Measure: Number; unit: percentage of participants
Arm/Group | Usual Care | FNPA Tool Intervention
Number analyzed (Participants) | 18 | 28
percentage of participants | 100 | 100

11. Secondary Outcome: BMI Z-score Change for Ages 4-10 Years
Time Frame: Baseline and 6 months post encounter
Measure: Mean (Standard Deviation); unit: BMI z-score
Arm/Group | Usual Care | FNPA Tool Intervention
Number analyzed (Participants) | 44 | 45
BMI z-score | 0.13 (0.69) | 0.04 (0.61)
Statistical Analysis 1: Comparison: Usual Care vs FNPA Tool Intervention; Test type: Superiority or Other; p = 0.4835, t-test, 2 sided

12. Secondary Outcome: BMI Z-score Change for Ages 11-17 Years
Time Frame: Baseline and 6 months post encounter
Measure: Mean (Standard Deviation); unit: BMI z-score
Arm/Group | Usual Care | FNPA Tool Intervention
Number analyzed (Participants) | 62 | 68
BMI z-score | 0.14 (0.32) | 0.11 (0.22)
Statistical Analysis 1: Comparison: Usual Care vs FNPA Tool Intervention; Test type: Superiority or Other; p = 0.5880, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from the date of initial encounter (enrollment date) to the date of the completion of the 6 month follow up survey data collection.
Arm/Group | Usual Care | FNPA Tool Intervention
Serious Adverse Events (participants affected / at risk) | 1/220 | 0/210
Other Adverse Events (participants affected / at risk) | 0/220 | 0/210
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Usual Care (N=220) | FNPA Tool Intervention (N=210)
Death of patient (Social circumstances) | 1 | 0 — One enrolled patient death occurred during the study period, however, the death was in no way related to participation in this research study. The patient's death occurred following 1 month data collection, but prior to the 6 month data collection.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No